CLINICAL TRIAL: NCT05156632
Title: A Multi-center, Randomized, Double-blind, Placebo-controlled Phase Ⅲb Clinical Trial to Evaluate the Efficacy, Immunogenicity and Safety of COVID-19 Vaccine (Vero Cell), Inactivated Booster Dose in Adults Aged 18 Years and Above
Brief Title: Efficacy,Immunogenicity and Safety of COVID-19 Vaccine , Inactivated Booster Dose in Adults Aged 18 Years and Above
Status: Withdrawn | Phase: Phase 3 | Type: Interventional
Why Stopped: The plan has changed
Sponsor: Sinovac Research and Development Co., Ltd. (Industry)
Responsible Party: Sponsor
Organization: Sinovac Biotech Co., Ltd (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: PRO-nCOV-3003
Record Dates: First submitted 2021-12-12; First posted 2021-12-14 (Actual); Last update posted 2023-02-08 (Actual); Status verified 2023-02

CONDITIONS: COVID-19
MeSH Terms: conditions — COVID-19 | interventions — sinovac COVID-19 vaccine; Aluminum Hydroxide

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Medium-dose group (Experimental): 4800 participants including 3400 participants aged 18-59 years ,1200 participants aged 60 years and above who have received 2 doses of CoronaVac® (medium-dose COVID-19 Vaccine) in an interval between 21-56 days will receive a booster dose of medium-dose COVID-19 Vaccine 5-8 months after their second dose.
  Interventions: Biological: Medium-dosage COVID-19 Vaccine,Inactivated
- High-dose group (Experimental): 4800 participants including 3400 participants aged 18-59 years,1200 participants aged 60 years and above who have received 2 doses of CoronaVac® (medium-dose COVID-19 Vaccine) in an interval between 21-56 days will receive a booster dose of high-dose COVID-19 Vaccine 5-8 months after their second dose.
  Interventions: Biological: High-dosage COVID-19 Vaccine,Inactivated
- Placebo group (Placebo Comparator): 4800 participants including 3400 participants aged 18-59 years,1200 participants aged 60 years and above who have received 2 doses of CoronaVac® (medium-dose COVID-19 Vaccine) in an interval between 21-56 days will receive a booster dose of placebo 5-8 months after their second dose.
  Interventions: Biological: Placebo-comparator group

INTERVENTIONS:
Biological: Medium-dosage COVID-19 Vaccine,Inactivated — The COVID-19 vaccine,inactivated was manufactured by Sinovac Research& Development Co., Ltd..600SU Inactivated SARS-COV-2 virus in 0·5 mL of aluminium hydroxide solution per injection.
  Other Names: Medium-dose CoronaVac®
  Arms: Medium-dose group
Biological: High-dosage COVID-19 Vaccine,Inactivated — The COVID-19 vaccine,inactivated was manufactured by Sinovac Research& Development Co., Ltd.1200SU inactivated virus in 0.5 mL of aluminium hydroxide solution per injection.
  Other Names: High-dose CoronaVac®
  Arms: High-dose group
Biological: Placebo-comparator group — The composition is aluminium hydroxide with no antigen ,0 SU/0.5 mL,The appearance of the placebo is consistent with the vaccine, which is a milky-white suspension.
  Other Names: Placebo (aluminum hydroxide)
  Arms: Placebo group

SUMMARY:
This is a multi-center, case-driven, randomized, double-blinded, and placebo-controlled Phase Ⅲb clinical trial of COVID-19 Vaccine manufactured by Sinovac Research & Development Co., Ltd.The purpose of this study is to evaluate the efficacy of the booster dose after two doses of CoronaVac® against RT-PCR confirmed symptomatic COVID-19 cases in participants aged 18 years and above.

DETAILED DESCRIPTION:
This is a multi-center, case-driven, randomized, double-blinded, and placebo-controlled Phase Ⅲb clinical trial of COVID-19 Vaccine manufactured by Sinovac Research & Development Co., Ltd.The purpose of this study is to evaluate the efficacy of the booster dose after two doses of CoronaVac® against RT-PCR confirmed symptomatic COVID-19 cases in participants aged 18 years and above.A total of 13,800 participants aged 18 years and above, who have received 2 doses CoronaVac® in an interval between 21-56 days will be enrolled.Participants will be enrolled and randomly assigned into 3 groups at a ratio of 1:1:1 to receive a booster dose of medium-dose or high-dose COVID-19 Vaccine or placebo 5-8 months after their second dose.Efficacy assessments will include the surveillance for COVID-19-like symptoms, the laboratory confirmation of SARS-CoV-2 infection by RT-PCR, and recording of COVID-19-related hospitalizations.All participants will be monitored for immediate reactions (within 30 minutes) after the booster dose vaccination, adverse events of special interest (AESIs) and serious adverse events (SAEs) for 6 months after booster dose inoculation. In addition,participants in reactogenicity subgroup will be monitored for local and systemic solicited adverse events (AEs) within 7 days and the unsolicited AEs within 28 days.Immunogenicity assessments will be determined by neutralizing and anti-SARS-CoV-2 S-protein antibodies in subgroup participants. The participants in the immunogenicity subgroup will be in the reactogenicity subgroup as well.

ELIGIBILITY:
Inclusion Criteria:

* Healthy adults aged 18 years and above, who have received 2 prior doses of CoronaVac® with an interval between those doses of 21-56 days, with the second dose given 5-8 months prior to the day of vaccination in the present study;
* The participants are able to understand and sign the informed consent voluntarily;
* Female participants who have a negative pregnancy test on the day of vaccination, and not currently breastfeeding;
* Must be willing to provide verifiable identification (in accordance with the local regulations), has means to be contacted and to contact the investigator during the study.

Exclusion Criteria:

* History of confirmed infection of SARS-CoV-2 prior to randomization;
* Any prior administration of another investigational coronavirus vaccine or current/planned simultaneous participation in another interventional study to prevent or treat COVID-19;
* Allergy to vaccines or vaccine/placebo ingredients, and serious adverse reactions to vaccines, such as urticaria, dyspnea, angioneurotic edema;
* Serious chronic disease, serious cardiovascular disease, hypertension and diabetes that cannot be controlled by drugs, hepatorenal disease, malignant tumor, etc;
* Acute central nervous system diseases such as encephalitis/myelitis, acute disseminating encephalomyelitis, and related disorders;
* Receipt of blood/plasma products or immunoglobulins in the past 3 months before vaccination;
* Participation in other studies involving study intervention within 30 days prior to vaccination;
* Receipt of attenuated live vaccines in the past 14 days prior to vaccination;
* Receipt of inactivated or subunit vaccines in the past 7 days prior to vaccination;
* Acute exacerbation or presentation of stable chronic diseases (including but not limited to asthma, migraine, gastrointestinal disorder, etc);
* Acute febrile illness with axillary temperature >37.5°C on the day of vaccination; enrollment could be considered if the fever is absent for 72 hours prior to vaccination;
* According to the investigator's judgment, the participant has any other factors that might interfere with the results of the clinical trial or pose additional risk to the participant due to participation in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2023-02-20 (Estimated); Primary Completion 2023-02-20 (Estimated); Study Completion 2023-02-20 (Estimated)

PRIMARY OUTCOMES:
Efficacy index -COVID-19 incidence | 6 months after booster dose
  COVID-19 incidence per 100 person-years of follow-up based on laboratory confirmed cases in participants aged 18 years and above, 6 months after booster dose

SECONDARY OUTCOMES:
Efficacy index -Confirmed hospitalized/severe/death incidence of COVID-19 | 6 months after booster dose
  Confirmed hospitalized/severe/death COVID-19 incidence per 100 person-years of follow-up based on laboratory confirmed cases, 6 months after booster dose
Safety index-Local reactions | Up to 7 days after booster dose
  Local reactions for up to 7 days after booster dose
Safety index-Systemic events | Up to 7 days after booster dose
  Systemic events for up to 7 days after booster dose
Safety index-AEs | Up to 28 days after booster dose
  AEs for up to 28 days after booster dose
Safety index-SAEs | Up to 6 months after booster dose
  SAEs for up to 6 months after booster dose

CONTACTS AND LOCATIONS:
Overall Officials: Javed Khan, Master, Principal Investigator — Rehman Medical Institute